CLINICAL TRIAL: NCT01991041
Title: European Registry of Anti-epileptic Drug Use in Patients With Lennox-Gastaut Syndrome (LGS).
Status: Completed | Type: Observational
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: E2080-E044-401
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Lennox-Gastaut Syndrome
Keywords: Lennox-Gastaut Syndrome
MeSH Terms: conditions — Lennox Gastaut Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Rufinamide
- Anti-Epileptic Drugs: Includes those used off label as part of local clinical practice

SUMMARY:
This is a registry study, where sites will enter patients with LGS who require a modification in anti-epileptic therapy (either the addition of another anti-epileptic drug, or the change of one drug to another). This will include patients who are started on rufinamide. Patients will be reviewed according to local practice, but it is envisaged that review will occur at approximately one month, three months and six months, and then every six months. Upon entry to the registry baseline details concerning disease severity, diagnosis, prior therapy, and developmental assessment will be recorded. On each subsequent visit the patient (usually through their caregiver) will be asked about current medication, general seizure profile, any seizures deemed to be of medical significance, tolerability, AEs (including suicidal-related events), and healthcare resource utilisation.

ELIGIBILITY:
INCLUSION CRITERIA

* Patients will be four years and older
* Patients will have an established diagnosis of Lennox-Gastaut syndrome, and:
* Documented history or current presence of multiple seizure types associated with LGS (including tonic or atonic seizures (drop attacks) and atypical absences)
* Documented history or current presence of typical EEG abnormalities (e.g., bursts of slow spike and wave activity)
* Presence of intellectual / learning disability (a variable degree is permitted)
* Patients entered on the registry will be those requiring a modification in their current anti-epileptic medication. This includes but is not limited to patients who are commenced on rufinamide as adjuvant therapy

EXCLUSION CRITERIA

* Female patients who are pregnant, lactating, or whom are planning to become pregnant
* Female patients, of child bearing potential, who are not willing to use appropriate contraception (This is at the discretion of the investigator)
* Those starting rufinamide and for whom the investigator considers it necessary to administer in contradiction to the indications, and warnings within the current Summary of Product Characteristics (SPC).

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participation in this study will be offered to any patient of four years or older, who has a known diagnosis of LGS, who requires a change in anti-epileptic therapy. This will include patients who are started on rufinamide, as an adjuvant therapy.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2008-06; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Safety during the use of rufinamide and other anti-epileptic drugs | At least three years
  Evaluation of the incidence of seizures of medical significance (including status epilepticus, new / worsening of seizure types and withdrawal seizures) during exposure to anti-epileptic drugs, including rufinamide, in patients with LGS; incidence of hypersensitivity reactions during the exposure to anti-epileptic drugs, including rufinamide; common AEs identified with anti-epileptic drugs, as they may be related to this specific population; including sedation, neurological AEs, suicidal-related events, events associated with blood dyscrasias, and the potential increased risk of infections.

SECONDARY OUTCOMES:
Long term use of rufinamide, and other anti-epileptic drugs | At least three years
  Evaluation, within the constraints of this population, of the impact on maturation anddevelopment that anti-epileptic drugs, including rufinamide, has on the LGS population; seizure control in LGS patients, including those taking rufinamide and other anti-epileptic drugs; assessment of healthcare resource utilisation.

CONTACTS AND LOCATIONS:
Locations (49):
- Austria (7):
  - Graz
  - Innsbruck
  - Linz
  - Mödling
  - Steyr
  - Vienna
  - Wein
- Denmark (2):
  - Copenhagen
  - Dianalund
- France (7):
  - Besançon
  - Lyon
  - Marseille
  - Paris
  - Reims
  - Strasbourg
  - Tain-l'Hermitage
- Germany (15):
  - Berlin
  - Bernau
  - Bielefeld
  - Bonn
  - Erlangen
  - Freiburg im Breisgau
  - Hamburg
  - Heidelberg
  - Jena
  - Kehl
  - Kiel
  - Münster
  - Stuttgart
  - Tübingen
  - Vogtareuth
- Italy (6):
  - Mantova
  - Milan
  - Padua
  - Roma
  - Trieste
  - Verona
- Spain (6):
  - Barcelona
  - Córdoba
  - Esplugues de Llobregat
  - Madrid
  - Málaga
  - Pamplona
- Lund, Sweden
- United Kingdom (5):
  - Birmingham
  - Cardiff
  - London
  - Manchester
  - West Yorkshire

REFERENCES:
- [Derived] Nikanorova M, Brandt C, Auvin S, McMurray R. Real-world data on rufinamide treatment in patients with Lennox-Gastaut syndrome: Results from a European noninterventional registry study. Epilepsy Behav. 2017 Nov;76:63-70. doi: 10.1016/j.yebeh.2017.08.026. Epub 2017 Sep 15. PMID 28927712